CLINICAL TRIAL: NCT06538961
Title: Immune Registry for BK (Polyomavirus Hominis 1) in Kidney Transplant Recipients
Brief Title: Immune Registry for BK in Kidney Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Other Study IDs: HM20028057
Record Dates: First submitted 2024-07-17; First posted 2024-08-06 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: BK Virus Infection; Kidney Transplant; Complications
Keywords: Immune Registry; BK in Kidney Transplant Recipients
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — 1. Biospecimens(blood) will be drawn for research purpose.
  2. Urine specimen collection
  Main study cohort:
  * specimen to assess BK-specific T cell immune responses will be collected at the time of transplant, 1 month, 2 month 3 month and 6 month post-transplant.
  * specimen to assess BK antibody responses will be collected at the time transplant, 3 month and 6 month post-transplant.
  * Uromap (urine gene expression test to detect for BK virus and rejection) will be performed on monthly basis for 6 months post-transplant in 10-18% of subjects.
  Sub-Study cohort:
  * specimen to assess BK-specific T cell immune responses and BK antibody responses will be collected on monthly basis for 6 month.
  * Uromap (urine gene expression test to detect for BK virus and rejection) will be performed on monthly basis for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Main study: Single organ deceased donor kidney transplant recipients. Main study group subjects are enrolled at the time of transplant.
  Interventions: Other: Blood samples: Main Study group; Other: Data Collection; Other: Urine Sample- Main Study group
- Sub-study: Single organ deceased donor Kidney Transplant Recipient who are newly diagnosed with BK Viremia or those with difficult-to-treat BKV > 3 logs (BKV log does not decrease by more than 1 log copy/ml drop on second per protocol lab). The sub-study group are enrolled once they are diagnosed with BK viremia post-transplant.
  Interventions: Other: Data Collection; Other: Urine sample- Sub-study group; Other: Blood sample: Sub-study group

INTERVENTIONS:
Other: Blood samples: Main Study group — the collection of blood samples at specified time points.
  Groups: Main study
Other: Data Collection — Donor and Recipient's clinical information including clinical history, demographic characteristics labs, and imaging.
Other: Urine Sample- Main Study group — -Post-transplant monthly urine sample collection for 6 months in 10-18% of subjects
  Groups: Main study
Other: Urine sample- Sub-study group — - Post-transplant monthly urine sample collection for 6 months in all subjects
  Groups: Sub-study
Other: Blood sample: Sub-study group — Monthly blood sample collection for 6 months
  Groups: Sub-study

SUMMARY:
Kidney transplantation (KT) is the best treatment modality available to date for patients with advanced kidney disease and the success of KT is dependent on maintaining a selective intricate balance between the risk of rejection and infections in KT recipients. BK virus is an important clinical infection affecting the post-transplant outcomes in KT recipients. BK nephropathy can affect 8-15% of patients after KT causing acute kidney injury, increased risk of rejection and fibrosis leading to additional hospital stays, increasing overall health care cost burden, and in some cases graft loss. The exact pathogenesis and treatment options for BK nephropathy are not clearly understood. It is debatable whether BK nephropathy is a full fledge donor-derived infection or reactivation of the recipient's latent infection. Irrespective of etiology, the common consensus is that treatment of BK virus infection depends on the selective restoration of host immune responses and balancing the risk of rejection vs worsening of infection.

DETAILED DESCRIPTION:
As with other viral infections, adaptive immunity plays an essential role in the control of BK virus infection. Previous studies have shown that humoral immunity doesn't prevent viral reactivation and cellular responses including CD4+ and CD8+ T cells play a crucial role in containing viral replication. Researchers have investigated the role of reconstitution of BK-specific T cell immunity KT recipients with overall low immunological risk populations showing that pre and post-transplant BK virus-specific cellular responses can be used as an important tool to identify KT recipients at increased risk of developing BK virus infection in the first year post-transplant. We plan to understand the role of adaptive immunity (cellular and humoral interplay) in a cohort with at least 50% of high immunological KT recipients with predominantly retransplant candidates, highly sensitized recipients with calculated panel reactive antibodies > 40 %, positive crossmatch or history of prior desensitization therapies.

The aim includes the sequential demonstration of immunogenesis processes that are specific to the BK virus in individuals who experience BK viremia and undergo various treatment approaches such as immunosuppression reduction and immune enhancement through intravenous immunoglobulins (IVIG).

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) male and female, deceased donor KT recipients
* Will include single organ transplants.
* Each participant must also have recently been diagnosed with BK viremia.
* In addition to the aforementioned inclusion criteria, each participant in the sub-study must also have recently been diagnosed with BK viremia or have difficult-to-treat BKV > 3 logs (BKV log does not decrease by more than 1 log copy/ml drop on second per protocol lab).

Exclusion Criteria:

* Prisoners will not be included in the study
* Multi-organ transplants and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults 18 and older who have undergone single organ deceased donor Kidney Transplant.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assessing the effect of kidney transplant immunosuppression therapy on the immune response against BK virus | 24 months
  Assessing the effect of kidney transplant induction and maintenance triple immunosuppression on humoral and cellular responses against BK virus compared at pre- and post-KT through clinical chart review, abnormal value or result from a clinical or laboratory evaluation, by assessing humoral and cellular responses against BK virus through BK specific T cell response, immunoglobulin G targeting BK levels, urine gene expression test to detect for BK virus and rejection.

SECONDARY OUTCOMES:
To identify the frequency risk of BK viremia | 24 month
  To identify the frequency risk of BK viremia post-transplant with careful monitoring of cellular and humoral responses against BK measured using BKV T cell immunity panel test, BKV IgG test, uromap(urine gene expression test to detect for BK virus and rejection), clinical chart review and abnormal values or results from a clinical laboratory evaluation including BKV PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Ambreen Azhar, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States